CLINICAL TRIAL: NCT06905028
Title: The Impact of Fasting on Disease Activity and the Gut Microbiota in Patients with Psoriasis and Psoriatic Arthritis - the RiseFast Pilot Study
Brief Title: Exploratory Clinical Study on Fasting in Psoriasis and Psoriatic Arthritis (RiseFast)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Max Delbrück Center for Molecular Medicine (MDC), Berlin (Unknown)
Responsible Party: Principal Investigator, Anika Rajput Khokhar, MD, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RiseFast
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Psoriasis Arthritis; Psoriasis (PsO)
Keywords: fasting; vegan; plant-based; diet; psoriasis
MeSH Terms: conditions — Psoriasis; Fasting | interventions — Diet, Plant-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fasting and Plant-Based Diet (Other): The participants (n=15 with PsO, n=15 with PsA) will undergo an initial 7-day fasting regime according to Buchinger (max. 350 kcal per day as liquids), followed by a dietary intervention that encompasses a plant-based diet (PBD) and time restricted eating (TRE) for 11 weeks.
  Interventions: Other: Fasting and Plant-Based Diet

INTERVENTIONS:
Other: Fasting and Plant-Based Diet — The participants will undergo an initial 7-day fasting regime according to Buchinger (max. 350 kcal per day as liquids), followed by a dietary intervention that encompasses a plant-based diet (PBD) and time restricted eating (TRE) for 11 weeks.

SUMMARY:
The RiseFast pilot study will investigate the clinical, metabolic and immunological effects of fasting and plant-based diet (PBD) on patients with psoriasis (PsO) and psoriatic arthritis (PsA) on their gut microbiota. The project will combine clinical assessments, cytometric profiling, and gut microbiota analysis to explore the relationship between fasting, a plant-based diet, and psoriatic disease. The study includes a 7-day fasting period followed by 11 weeks of PBD, with the goal of improving disease activity, quality of life, and understanding the role of gut microbiota in these conditions. This approach could lead to low-cost, accessible therapeutic options with minimal side effects.

DETAILED DESCRIPTION:
Psoriatic disease, encompassing psoriasis (PsO) and psoriatic arthritis (PsA) is a chronic inflammatory condition influenced by genetic, immune, and environmental factors, particularly diet and gut microbiota. While biologics and DMARDs have improved disease management, treatment responses vary, and long-term remission remains difficult. Continuous inflammation control often requires pharmacological treatment, highlighting the need for adjunctive therapies.

Emerging research links gut microbiota imbalances (dysbiosis) to chronic inflammation, suggesting that dietary interventions could offer therapeutic benefits. Fasting and plant-based diets (PBD) may help regulate immune responses and gut microbiota composition. Fasting has been shown to reduce oxidative stress, promote autophagy, and alter immune cell dynamics, while PBD is associated with anti-inflammatory effects and enhanced microbial diversity.

The RiseFast Pilot Study aims to investigate whether a seven-day fasting period followed by a structured PBD can improve disease activity, quality of life, and gut microbiota in PsO and PsA patients. While prior studies suggest potential benefits, their specific effects on psoriatic disease remain unclear. By integrating clinical, microbiome, and immune profiling, the study aims to clarify dietary impacts on inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Active plaque psoriasis (PASI ≥3) or Psoriatic Arthritis fulfilling the Classification Criteria for Psoriatic Arthritis (CASPAR) and not meeting MDA criteria
* on stable baseline psoriatic treatment for 12 weeks before enrollment
* ≥ 18 years old

Exclusion Criteria:

* Pregnancy or breastfeeding
* underweight (BMI ≤18,5)
* eating disorder in the last 5 years
* severe internal diseases (e.g. renal insufficiency with creatinine > 2mg/dl)
* current practice of vegan diet or fasting within the past 6 months
* use of antibiotics within the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Changes in disease activity measured by the Psoriasis Area and Severity Index (PASI) after 12 weeks compared to baseline.
Disease Activity index for PSoriatic Arthritis (DAPSA) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Changes in disease activity measured by the Disease Activity index for Psoriatic Arthritis (DAPSA) after 12 weeks compared to baseline.

SECONDARY OUTCOMES:
Sociodemographic Measurements | Date of inclusion (baseline)
  age, education level, household income, employment status, marital status, complete family history of Psoriasis and/or Psoriatic Arthritis in first- and second-degree relatives, current and previous illness and co-morbidities, and current medications.
Medication intake | Date of inclusion (baseline), after 6 and 12 weeks
  Systematized documentation of medication, main and secondary diagnoses using CRF.
Quantification of Behavioral Factors | Date of inclusion (baseline), after 6 and 12 weeks
  Sleeping habits, Physical Activity, Stress and Media Consumption via Likert Scales, range from 0 to 10 while higher values meaning a higher grade of agreement.
Behavioral Factors: alcohol consumption | Date of inclusion (baseline), after 6 and 12 weeks
  Number of alcoholic beverages on average per week in the last month.
Behavioral Factors: smoking | Date of inclusion (baseline), after 6 and 12 weeks
  Smoking status in packyears.
Expectation questions | Date of inclusion (baseline)
  For fasting on a 10-point likert scale from 1 (nothing at all) to 10 (very strong).
Resting blood pressure (mmHg) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
Pulse rate (bmp) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
Abdominal circumference (cm) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
Waist to Hip Ratio (cm) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
Weight (kg) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Change in weight (kg)
Body Mass Index (kg/m2) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Change in Body Mass Index measured as weight (kg) and height (m) (kg/m^2)
Bio-electrical impedance analysis (BIA) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Estimation of the body composition via bio-electrical impedance analysis (body fat and visceral fat in %)
Body Surface Area (BSA) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Body Surface Area (BSA) quantifies the percentage of skin affected by psoriasis, with one palm equating to approximately 1% of the total body surface. Values range from 0% to 100%, with higher percentages indicating greater skin involvement.
Nail Psoriasis Severity Index (NAPSI) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Nail Psoriasis Severity Index (NAPSI) evaluates the severity of nail psoriasis. It assesses each fingernail for specific features in the nail matrix (pitting, leukonychia, crumbling, red spots in the lunula) and nail bed (onycholysis, splinter hemorrhages, subungual hyperkeratosis, oil drop discoloration). Each nail is scored from 0 to 8, with higher scores indicating more severe nail involvement.
Criteria of minimal disease activity (MDA) or very low disease activity (VLDA) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Minimal Disease Activity (MDA) is a composite assessment of disease activity state in PsA. It includes 7 components: tender joint count (68) ≤ 1, swollen joint count (66) ≤ 1, Psoriasis Area Severity Index ≤ 1/Body Surface Area ≤ 3, enthesitis≤ 1, patient global assessment of disease activity VAS ≤ 20, pain VAS ≤ 15 and HAQ-DI ≤ 0.5. MDA requires 5 out of 7 components to be met
  Very Low Disease Activity (VLDA) is a stricter composite assessment of disease activity state in Psoriatic Arthritis (PsA). It includes 7 components, all of which must be fulfilled to achieve VLDA: tender joint count (68): ≤ 1; Swollen joint count (66): ≤ 1; Psoriasis Area and Severity Index (PASI): ≤ 1 or Body Surface Area (BSA): ≤ 1%; Enthesitis count: 0 (no active enthesitis); Patient global assessment of disease activity (VAS): ≤ 20; Pain assessment (VAS): ≤ 15; Health Assessment Questionnaire Disability Index (HAQ-DI): ≤ 0.5
68 Tender Joint Count | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Change in Tender Joint Count at Week 12 as compared to baseline, with a maximum possible range between 0 to 68 with higher values indicating a worsening of the symptoms.
66 Swollen Joint Count | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Change in Swollen Joint Count at Week 12 as compared to baseline, with a maximum possible range between 0 to 66 with higher values indicating a worsening of the symptoms.
Leeds Enthesitis Index (LEI) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Leeds Enthesitis Index (LEI) is used to assess enthesitis in psoriatic arthritis (PsA). It evaluates tenderness (1 = present, 0 = absent) at six specific sites: the lateral epicondyles (elbows), medial femoral condyles (knees), and Achilles tendon insertions (heels) on both sides of the body. The total score ranges from 0 (no tenderness) to 6 (tenderness at all sites).
ACR20/50 criteria | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  ACR20/50 and ACR50 response criteria assess treatment efficacy in psoriatic arthritis. Achievement of ACR20 requires a ≥20% improvement in both the tender joint count (68 joints) and the swollen joint count (66 joints), in addition to a ≥20% improvement in at least three of the following five domains: patient global assessment of disease activity (VAS 0-100), physician global assessment of disease activity (VAS 0-100), pain assessment (VAS 0-100), physical function (e.g., HAQ-DI), and acute-phase reactants (CRP or ESR). Similarly, ACR50 requires a ≥50% improvement in these parameters, reflecting a more substantial reduction in disease activity.
Health Assessment Questionnaire Disability Index (HAQ-DI) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Change from Baseline in the HAQ after 12 weeks, range from 0 to 3 while higher values meaning a higher grade of disability.
Quality of Life questionnaire (WHO-5) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Change from Baseline in the WHO-5, range from 0 to 100 %, higher values meaning a higher grade of well-being.
Dermatology Life Quality Index (DLQI) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Changes from Baseline in the DLQI after 12 weeks, range from 0 to 3, higher values meaning a lower grade of life quality.
EULAR Psoriatic Arthritis Impact of Disease (PsAID12) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Changes from Baseline in the PsAID-12, formed of 12 questions, each evaluated on a 0-10 numeric rating scale, where a higher score reflects a greater impact of PsA.
Subjective strength of the main complaint (Visual Analogue Scale) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  The Visual Analog Scale for Pain (VAS Pain) and the Visual Analog Scale for Skin Complaints (VAS Skin Complaints) both range from 0 to 10, with higher values indicating more severe symptoms.
Short Form 36 | Date of inclusion (baseline) and after 12 weeks
  36-Item Short Form Survey (SF-36) used as Quality of life assessment, containing 36 items, the total score range from 0 to 100, a high score represents a high quality of life).
Food selection | Date of inclusion (baseline), after 4 and 9 weeks
  Nutritional history via dietary record (3-day food record)
Dietary Behaviour | Date of inclusion (baseline), after 6 and 12 weeks
  The Food Frequency Questionnaire (FFQ) records dietary behaviors such as mealtimes, frequency of food intake, food preferences, and fasting experiences.
Differential blood count | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Analysis of different types of blood cells to assess immune status and detect possible infections or inflammations.
CRP in milligram per liter (mg/L) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  CRP (C-reactive protein) as a marker of inflammatory conditions is used to assess acute inflammation and monitor the effects of prolonged fasting and plant-based nutrition. Higher scores indicate more inflammation.
Creatinine in µmol per liter (µmol/L) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Biomarker of renal function and muscle metabolism.
Ketone bodies (mmol/l) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Indicators of fat metabolism and ketosis, analyzed for metabolic adaptations.
Glucose (mg/dl) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Fasting blood sugar measurement to monitor metabolic changes.
Hepatic transaminases (ALAT, ASAT) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  * ALAT in units per liter (U/L)
  * ASAT (U/L)
Electrolytes | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  * calcium in millimol per liter (mmol/L)
  * potassium (mmol/L)
  * sodium (mmol/L)
Flow cytometry: Phenotyping of immune cells | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Determination of cytometric parameters to assess changes in cell activation and quantify alterations in the absolute and/or relative sizes of immune cell subpopulations (e.g., classical, intermediate, and non-classical monocytes; naïve and memory T-cells; B-cell differentiation to plasmablasts and plasma cells). In addition, gene expression analysis of immune cells using Affymetrix whole genome microarrays and RNA sequencing (RNAseq) will be conducted to explore transcriptional patterns and identify markers that could reveal relevant immune cell subpopulations, which are not yet captured in the cytometric phenotyping screen.
Cytokine profile | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Quantification of pro- and anti-inflammatory cytokines (e.g., IL-6, IL-17, TNF-α, IL-10) using multiplex ELISA or Luminex technology.
Functional immune cell tests | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Ex vivo stimulation of immune cells to measure proliferation capacity and cytokine secretion.
NK cell activity | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Determination of cytotoxic function of natural killer (NK) cells.
Autoantibodies | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Screening for disease-relevant autoantibodies associated with immune dysregulation.
Gene expression analysis | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  RNA sequencing of whole blood samples to assess diet-induced transcriptomic changes.
Epigenetic analysis | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  DNA methylation profiling to examine nutrition-related epigenetic modifications.
Metabolomics | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Targeted and untargeted metabolite profiling of energy, lipid, and amino acid metabolism.
Biobanking (for future proteomics analysis) | Date of inclusion (baseline), day 8, after 6 and 12 weeks
  Sample storage for additional protein analysis if funding is secured.
Gut microbiota characterization | Date of inclusion (baseline), day 8 or first stool after fasting, after 6 and 12 weeks
  Molecular profiling of the highly individualized intestinal microbiota composition is performed through 16S rDNA gene sequencing of stool samples, aiming to identify fasting- and diet-induced alterations in the gut microbiota.

OTHER OUTCOMES:
Final questionnaire to record tolerability of fasting and nutrition, adverse effects | After 12 weeks
  Measurement of tolerability of fasting and nutrition as well as adverse effects via Likert Scales, range from 0 to 10 while higher values meaning a higher grade of agreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Charité - Universitätsmedizin Berlin, Psoriasis-Forschungs- und BehandlungsCentrum, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No